CLINICAL TRIAL: NCT02207296
Title: Operative Hemodynamic Optimization Using the Plethysmographic Variability Index During Orthopedic Surgery : a Multicentric Prospective Randomized Controlled Study
Brief Title: Operative Hemodynamic Optimization Using the Plethysmographic Variability Index During Orthopedic Surgery
Acronym: OPVI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-A00330-47
Record Dates: First submitted 2014-06-17; First posted 2014-08-04 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Hip Arthroplasty; Knee Arthroplasty; General Anesthesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- PVI group (Other): Fluid optimisation using PVI
  Interventions: Device: Plethysmographic variability index
- Control group (No Intervention): Standard care using a hemodynamic protocol during general anesthesia

INTERVENTIONS:
Device: Plethysmographic variability index
  Arms: PVI group

SUMMARY:
The purpose of this study is to determine whether an operative hemodynamic optimization using the plethysmographic variability index during orthopedic surgery could decrease the length of hospital stay and the postoperative morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Indication to a knee or hip arthroplasty under general anesthesia
* Sinusal rhythm

Non Inclusion Criteria:

* Pregnant women
* Black skin
* Dialysis
* Cardiac arrythmia
* Sepsis
* Use of another hemodynamic monitoring during surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay after knee or hip arthroplasty | Real length of hospital stay expressed as number of day (maximum 60 days)
  Surgeons, blinded to the group allocation, are the postoperative care providers who decide the length of hospital stay.

SECONDARY OUTCOMES:
Troponin value | Postoperative Day 1 and Day 3
Creatinine value | Postoperative Day 1 and Day 3
Arterial Lactate | 1 hour after end of surgery
Postoperative cardiac complications | Participants will be followed for the duration of hospital stay, an expected average of 1 week, until postoperative day 60
Theorical length of hospital stay after knee or hip arthroplasty | Theorical length of hospital stay expressed as number of day (maximum 60 days)
  Evaluation twice per day starting day 3 until up day 60. A check list was used by an independant investigator to define the theorical date of end hospitalisation, from day 3 until day 60

OTHER OUTCOMES:
Medico economic evaluation | Participants will be followed for the duration of hospital stay, an expected average of 1 week, until postoperative day 60

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France

REFERENCES:
- [Derived] Fischer MO, Daccache G, Lemoine S, Tavernier B, Compere V, Hulet C, Bouchakour CE, Canevet C, Gerard JL, Guittet L, Lorne E, Hanouz JL, Parienti JJ. The OPVI trial - perioperative hemodynamic optimization using the plethysmographic variability index in orthopedic surgery: study protocol for a multicenter randomized controlled trial. Trials. 2015 Nov 4;16:503. doi: 10.1186/s13063-015-1020-7. PMID 26537815